CLINICAL TRIAL: NCT03301779
Title: Clinical Investigation to Evaluate the New Health Sciences Hemanext® Oxygen Reduction System for Leukoreduced Red Blood Cells With CP2D Anticoagulant and AS-3 Additive - Pivotal Trial
Brief Title: Clinical Investigation to Evaluate the Hemanext® Oxygen Reduction System - Pivotal Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hemanext (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CLIN-0001
Record Dates: First submitted 2017-09-25; First posted 2017-10-04 (Actual); Results first posted 2020-03-17 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Whole Blood Donation and Leukoreduction
Keywords: Red Blood Cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Investigational Product (Experimental): Blood product from these donors will be processed and stored using the Hemanext Red Blood Cell Processing System
  Interventions: Device: Hemanext Red Blood Cell Processing System
- Control Product (No Intervention): Blood product from these donors will be stored in a Haemonetics Leukotrap Whole Blood System.

INTERVENTIONS:
Device: Hemanext Red Blood Cell Processing System — Leukoreduced red blood cell product from donors in the Investigational Product arm will be processed in the Hemanext Oxygen Reduction Bag for 3 hours and then transferred to the Hemanext Storage Bag and stored for 42 days at 1-6°C.
  Arms: Investigational Product

SUMMARY:
The primary goal of Hemanext. is to improve red cell storage through novel storage methods. Based on our review of the pertinent literature, there is substantial evidence suggesting that prolonged exposure to oxygen during storage results in oxidative damage to the red blood cells leading to decreased therapeutic potential. Therefore, removal of oxygen from red blood cell products prior to storage has potential to preserve the cells in a more physiologically relevant state.

Currently, Hemanext has focused on the design and development of a dual compartment bag system designated as the Hemanext Red Blood Cell Processing System. After standard processing of donated whole blood units into leukoreduced packed red blood cells (LR-RBCs) with the appropriate additive solutions, the LR-RBCs would then be placed in the oxygen reduction bag (ORB) which allows for the rapid diffusion of oxygen out of the blood, through a sterile, oxygen-permeable membrane, and into iron-based oxygen sorbents. After processing, the blood is transferred again from the ORB into the Hemanext storage bag (HSB) which will preserve the anaerobic state of the LR-RBC product for the duration of cold storage.

Hemanext has conducted preliminary storage tests to ascertain the effects of anaerobic storage on overall blood health in various storage solutions. The research team has focused primarily on percent hemolysis, which is mandated by the FDA to remain below 1% for the duration of storage, as well as ATP and 2,3-DPG levels.

DETAILED DESCRIPTION:
In vitro and in vivo performance of O2/CO2 reduced red blood cells produced with the Hemanext System will be used to demonstrate the acceptability the final product for clearance. To accomplish this, the study will require a total of 100 studyevaluable donors. completing the study. The study entails a randomized, paired, 2-x-2 crossover design where every study donor (n = 10093) evaluable study donors who completes the study will donate a total of two whole blood units with individual units being donated at least 56 days (8 weeks) apart. One unit will be used as the test and the other unit will be used for the control. The order in which the IP and the CP will be used to collect, filter and store the whole blood and appropriate blood products (within the context of the crossover design) will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Study donor must be ≥ 18 years of age.
* Study donor must be ≥ 110 pounds.
* Study donor's body temperature must be ≤ 37.5°C / 99.5°F (oral).
* Study donor's hemoglobin must be ≥12.5 g/dL if female and ≥13.0 g/dL if male.
* Study donor's hematocrit must be ≥ 38% if female and ≥39% if male.Study participants must meet EITHER hemoglobin or hematocrit criteria.
* Study donor must meet all criteria per respective site's Research Blood Donation Record (BDR).
* Study donor's most recent single RBC unit donation must have been ≥56 days prior to study donation.
* Study donor's most recent double RBC unit donation must have been ≥ 112 days prior to study donation.
* Study donor must have consented to study participation by reviewing and having expressed understanding the site-respective IRB-approved informed consent form prior to undergoing any study related procedures.

  21 CFR 50
* Study donor's testing results from collected blood does not indicate a risk of transfusion-transmitted disease (TTD)*.
* Study donors must agree to report adverse events from the time of signing the informed consent to twenty-four hours following the end of their active study involvement.
* Female study donors must not be pregnant, expected to be pregnant or breastfeeding.
* Female donors who participate in the in vivo portion of the study:

Women of child-bearing age must not be pregnant as determined by a negative pregnancy test prior to each re-infusion. If acceptable by local procedures, post-menopausal or surgically sterile women may be exempt from the pregnancy testing requirement.

Exclusion Criteria:

* Study donor is < 18 years of age.
* Study donor < 110 pounds.
* Study donor's body temperature is > 37.5°C / 99.5°F (oral).
* Study donor's hemoglobin is < 12.5 g/dL if female and < 13.0 g/dL if male.
* Study donor's hematocrit is < 38% if female and < 39% if male.
* Study donor does not meet all criteria per respective site's Research Blood Donation Record (BDR).
* Study donor's most recent single RBC unit donation was < 56 days prior to study donation.
* Study donor's most recent double RBC unit donation was < 112 days prior to study donation.
* Study donor has not consented to study participation.
* Study donor's testing results from collected blood does indicate a risk of transfusion-transmitted disease (TTD)*.
* Female donors who participate in the in vivo portion of the study: study donor is pregnant, expected to be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faye West, MD, Principal Investigator — American Red Cross Mid-Atlantic Research Facility; Jose A Cancelas Perez, MD, PhD, Principal Investigator — Hoxworth Blood Center; Matthew Karafin, MD, Principal Investigator — Versiti Blood Health
Locations (3):
- United States (3):
  - Hoxworth Blood Center, University of Cincinnati, Cincinnati, Ohio
  - American Red Cross Mid-Atlantic Research Facility, Norfolk, Virginia
  - Blood Center of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were immediately assigned to a group upon enrollment.
Groups:
- Investigational Product First, Then Control Product: A donor randomized to this arm donated their first whole blood unit to be stored with the Investigational Product.These units were processed in the Hemanext Oxygen Reduction Bag for 3 hours and then transferred to the Hemanext Storage Bag and stored for 42 days at 1-6°C.
  These donors then donated their second whole blood unit to be stored with the Control Product. These units were stored in a Haemonetics Leukotrap Whole Blood System for 42 days at 1-6°C.
- Control Product First, Then Investigational Product: A donor randomized to this arm donated their first whole blood unit to be stored with the Control Product. These units were stored in a Haemonetics Leukotrap Whole Blood System for 42 days at 1-6°C.
  These donors then donated their second whole blood unit to be stored with the Investigational Product.These units were processed in the Hemanext Oxygen Reduction Bag for 3 hours and then transferred to the Hemanext Storage Bag and stored for 42 days at 1-6°C.
Period: Overall Study
Arm/Group | Investigational Product First, Then Control Product | Control Product First, Then Investigational Product
Started | 48 | 52
Completed | 40 | 45
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- All Study Donors: This study was a crossover design and all Donors donated units to both the Investigation and Control arms so the Baseline Measures for all donors are combined here irrespective of their randomization.
Arm/Group | All Study Donors
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 98
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 10
  White | 88
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: % of Red Blood Cells With Hemolysis
Description: Percentage of packed Red Blood Cell units with hemolysis at day 42 of storage.
Time Frame: On day 42 of storage
Measure: Mean (Standard Deviation); unit: % of Red Blood Cells with Hemolysis
Groups:
- Investigational Product: Blood products from these donors will be processed and stored using the Hemanext Red Blood Cell Processing System.
  Hemanext Red Blood Cell Processing System: Leukoreduced red blood cell product from donors in the Investigational Product arm will be processed in the Hemanext Oxygen Reduction Bag for 3 hours and then transferred to the Hemanext Storage Bag and stored for 42 days at 1-6°C.
- Control Product: Blood products from these donors will be stored in a Haemonetics Leukotrap Whole Blood System.
Arm/Group | Investigational Product | Control Product
Number analyzed (Participants) | 95 | 94
% of Red Blood Cells with Hemolysis | 0.29 (0.168) | 0.29 (0.152)

2. Primary Outcome: Dual Label 24 Hour In Vivo % Recovery of Red Blood Cells
Description: The mean 24-hour, post-transfusion, in vivo red blood cell recovery.
Time Frame: Day 42 of storage
Measure: Mean (Standard Deviation); unit: % Recovery of Red Blood Cells
Arm/Group | Investigational Product | Control Product
Number analyzed (Participants) | 19 | 21
% Recovery of Red Blood Cells | 89.3 (5.81) | 85.8 (6.12)

3. Primary Outcome: % Red Blood Cells Recovered Post-Filtration
Description: Percentage of red blood cells recovered after the filtration process.
Time Frame: Post-Filtration on Day 0
Measure: Mean (Standard Deviation); unit: % of Red Blood Cells Recovered
Arm/Group | Investigational Product | Control Product
Number analyzed (Participants) | 98 | 96
% of Red Blood Cells Recovered | 92.3 (1.9) | 91.1 (4.31)

ADVERSE EVENTS:
Time Frame: Study-related adverse events are defined as those study participant-reported adverse events occurring within 24-hours of donation and/or transfusion. Non-study-related adverse events outside of these periods were not recorded unless they were of a nature to impact study participant evaluability, safety or data validity.
Arm/Group | Investigational Product | Control Product
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 1/100 | 1/100
Other Adverse Events (participants affected / at risk) | 9/100 | 9/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Product (N=100) | Control Product (N=100)
Appendicits (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Product (N=100) | Control Product (N=100)
Subject called to say he had dizziness at work after donation. (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dizzyness after donation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Light-headedness after donation (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Bruising or pain on arm at blood donation site (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Nausea after donation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cardiac Ablation (Cardiac disorders) | 1 (1) | 1 (1) — Participant had the procedure during their participation in the study so it was recorded as an adverse event.
Side Pain (Infections and infestations) | 1 (1) | 1 (1) — This adverse event caused the participant to go see their primary care physician and lead to the discovery that they had appendicitis (recorded in the serious adverse event section)

LIMITATIONS AND CAVEATS:
Disclaimer: The 51-Cr/99-Tc(m) labeling for 14 study subjects occurred without prior RDRC approval and was done at a site that did not meet GMP standards.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03301779/Prot_SAP_000.pdf